CLINICAL TRIAL: NCT00196716
Title: A Multicenter, Open-label Study of Low Dose Maintenance Treatment of Fabrazyme (Recombinant Human Alpha-Galactosidase A (R-h Alpha-GAL)) Replacement Therapy in Patients With Fabry Disease
Brief Title: A Study of the Safety and Efficacy of Fabrazyme in Patients With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL-017-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2009-04-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Fabry Disease
Keywords: alpha Galactosidase A; aGAL; rh aGAL; Fabry; GL3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

ARMS (1):
- Fabrazyme (Experimental): Open-label study. Patients received 1.0 mg/kg Fabrazyme every two weeks for approximately six months followed by 0.3 mg/kg Fabrazyme every two weeks for approximately 18 months.
  Interventions: Biological: Fabrazyme (agalsidase beta)

INTERVENTIONS:
Biological: Fabrazyme (agalsidase beta) — 1.0 mg/kg Fabrazyme every two weeks for approximately six months followed by 0.3 mg/kg Fabrazyme every two weeks for approximately 18 months
  Other Names: r-hαGAL

SUMMARY:
People with Fabry disease have an alteration in their genetic material (DNA) which causes a deficiency of the alpha-galactosidase A enzyme. This enzyme helps to break down and remove certain types of fatty substances called "glycolipids." These glycolipids are normally present within the body in most cells. In people with Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because alpha-galactosidase A is not present, or is present in small quantities. The build up of glycolipid levels (also referred to as "globotriaosylceramide" or "GL-3") in these tissues is thought to cause the clinical symptoms that are common to Fabry disease. Symptoms commonly appear during childhood with pain in the hands and feet. This trial is designed to evaluate the efficacy of a lower dose of Fabrazyme in patients who initially received 1.0 mg/kg every 2 weeks of Fabrazyme by investigating if the achieved clearance of glycosphingolipid deposits in the vascular endothelium of the kidney can be maintained at a lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Have clinical manifestations of Fabry disease
* All patients have to have a plasma αGAL activity of < 1.5 nmol/hr/mL or a documented leukocyte αGAL activity of < 4 nmol/hr/mg
* Patient or patient's parent/guardian had to provide written informed consent prior to any study-related procedures being performed
* Patients had to be male and ≥ 16 years of age

Exclusion Criteria:

* There is evidence of renal insufficiency, as defined by serum creatinine greater than or equal to 2.2 mg/dL (194.7 μmol/L) AND/OR has an estimated glomerular filtration rate (GFR) of <80 mL/min (using the equation derived from the Modification of Diet in Renal Disease Study (MDRD))
* Has undergone kidney transplantation or is currently on dialysis
* Has a clinically significant organic disease or an unstable condition (with the exception of symptoms relating to Fabry disease) that in the opinion of the Investigator would preclude participation in the trial
* Has participated in a study employing an investigational drug within 30 days of the start of this trial
* Patients who received prior treatment with enzyme replacement therapy for Fabry disease
* Patient was unable to comply with the requirements of the protocol

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-06; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (4):
- II. interní klinika 1. LF UK, Prague, Czechia
- Tartu University Clinics, Department of Internal Medicine, Tartu, Estonia
- Klinika Chorob Metabolicznych, Instytut "Pomnik-Centrum Zdrowia Dziecka", Warsaw, Poland
- Detská fakultná nemocnica Kramáre I. Interná klinika, Bratislava, Slovakia

RESULTS

PARTICIPANT FLOW:
Period: 1.0 mg/kg Period
Arm/Group | Fabrazyme
Started | 21
Completed | 21
Not Completed | 0
Period: 0.3 mg/kg Period
Arm/Group | Fabrazyme
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 21

OUTCOME MEASURES:

1. Primary Outcome: Globotriaosylceramide (GL-3) Clearance in Kidney Interstitial Capillary Endothelium
Description: Kidney biopsies were taken at Baseline, Week 24, and Week 96 and analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Each biopsy was evaluated by pathologists for the total number of vessels with GL-3 accumulation on an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe).
Time Frame: Throughout study; 96 weeks
Population: Intent-to-Treat (ITT) Population. One patient switched back to 1.0 mg/kg Fabrazyme treatment at Week 76 and therefore assessments at Week 76 and thereafter for this patient were excluded from the analysis.
Measure: Number; unit: Participants
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
Participants
  Zero (0) Kidney GL-3 Score at Baseline | 3
  Zero (0) Kidney GL-3 Score at Week 24 | 21
  Zero (0) Kidney GL-3 Score at Week 96 | 18
  Mild (1) Kidney GL-3 Score at Baseline | 17
  Mild (1) Kidney GL-3 Score at Week 24 | 0
  Mild (1) Kidney GL-3 Score at Week 96 | 2
  Moderate (2) Kidney GL-3 Score at Baseline | 1
  Moderate (2) Kidney GL-3 Score at Week 24 | 0
  Moderate (2) Kidney GL-3 Score at Week 96 | 0
  Severe (3) Kidney GL-3 Score at Baseline | 0
  Severe (3) Kidney GL-3 Score at Week 24 | 0
  Severe (3) Kidney GL-3 Score at Week 96 | 0

2. Secondary Outcome: Skin Globotriaosylceramide (GL-3) Clearance From Superficial Skin Capillary Endothelium
Description: Skin biopsies were taken at Baseline, Week 24, Week 48, Week 72, and Week 96 and analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Each biopsy was evaluated by pathologists for the total number of vessels with GL-3 accumulation on an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe).
Time Frame: Throughout study ; 96 weeks
Population: ITT Population. One patient switched back to 1.0 mg/kg Fabrazyme treatment at Week 76 and therefore assessments at Week 76 and thereafter for this patient were excluded from the analysis.
Measure: Number; unit: Participants
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
Participants
  Zero (0) Skin GL-3 Score at Baseline | 5
  Zero (0) Skin GL-3 Score at Week 24 | 20
  Zero (0) Skin GL-3 Score at Week 48 | 15
  Zero (0) Skin GL-3 Score at Week 72 | 17
  Zero (0) Skin GL-3 Score at Week 96 | 16
  Mild (1) Skin GL-3 Score at Baseline | 1
  Mild (1) Skin GL-3 Score at Week 24 | 1
  Mild (1) Skin GL-3 Score at Week 48 | 4
  Mild (1) Skin GL-3 Score at Week 72 | 3
  Mild (1) Skin GL-3 Score at Week 96 | 2
  Moderate (2) Skin GL-3 Score at Baseline | 11
  Moderate (2) Skin GL-3 Score at Week 24 | 0
  Moderate (2) Skin GL-3 Score at Week 48 | 2
  Moderate (2) Skin GL-3 Score at Week 72 | 1
  Moderate (2) Skin GL-3 Score at Week 96 | 2
  Severe (3) Skin GL-3 Score at Baseline | 4
  Severe (3) Skin GL-3 Score at Week 24 | 0
  Severe (3) Skin GL-3 Score at Week 48 | 0
  Severe (3) Skin GL-3 Score at Week 72 | 0
  Severe (3) Skin GL-3 Score at Week 96 | 0

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Evaluated at Baseline, Week 24 and Week 96. eGFR is an estimation of the glomerular filtration rate of the kidneys (how much blood the kidneys are filtering). For this study, normal eGFR was defined as greater than 90 mL/min/1.73 m2
Time Frame: Throughout study; 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m2
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
ml/min/1.73 m2
  eGFR at Baseline | 92.5 (21.12) [2 to 7]
  eGFR at Week 24 | 93.1 (24.10)
  eGFR at Week 96 | 92.8 (27.42)

4. Secondary Outcome: Plasma Globotriaosylceramide (GL-3)
Description: Evaluated at Baseline, Week 24, Week 48, Week 72 and Week 96. Plasma GL-3 is often elevated in the plasma of patients diagnosed with Fabry disease. This outcome measure evaluated the mean plasma GL-3 values for all patients to see if it decreased while on Fabrazyme. Normal plasma GL-3 level was <= 7.03 µg/mL.
Time Frame: Throughout study; 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
μg/mL
  Plasma GL-3 values at Baseline | 12.24 (3.369)
  Plasma GL-3 values at Week 24 | 5.18 (1.276)
  Plasma GL-3 values at Week 48 | 5.50 (1.480)
  Plasma GL-3 values at Week 72 | 5.64 (1.635)
  Plasma GL-3 values at Week 96 | 6.53 (1.497)

5. Secondary Outcome: Urine Globotriaosylceramide (GL-3)
Description: Evaluated at Baseline, Week 24 and Week 96. Urine GL-3 is often elevated in the urine of patients diagnosed with Fabry disease. This outcome measure evaluated the mean urine GL-3 in first morning void urine for all patients to see if it decreased while on Fabrazyme. Normal Urine GL-3 threshold was < 8.8 μg/mg.
Time Frame: Throughout study, 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mg
Arm/Group | Fabrazyme
Number analyzed (Participants) | 21
μg/mg
  Urine GL-3 values at Baseline | 221.3 (152.0)
  Urine GL-3 values at Week 24 | 109.2 (120.00)
  Urine GL-3 values at Week 96 | 122.5 (181.06)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- 1.0 mg/kg Fabrazyme: 1.0 mg/kg Fabrazyme, Week 0 to Week 24.
- 0.3 mg/kg Fabrazyme: 0.3 mg/kg Fabrazyme, Week 24 to Week 96.
Arm/Group | 1.0 mg/kg Fabrazyme | 0.3 mg/kg Fabrazyme | Total
Serious Adverse Events (participants affected / at risk) | 0/21 | 4/21 | 5/21
Other Adverse Events (participants affected / at risk) | 9/21 | 12/21 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.0 mg/kg Fabrazyme (N=21) | 0.3 mg/kg Fabrazyme (N=21) | Total (N=21)
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.0 mg/kg Fabrazyme (N=21) | 0.3 mg/kg Fabrazyme (N=21) | Total (N=21)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 2 | 0 | 2
Ventricular hypertrophy (Cardiac disorders) | 0 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 4
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chills (General disorders) | 3 | 1 | 3
Fatigue (General disorders) | 0 | 1 | 1
Feeling abnormal (General disorders) | 1 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 3
Bronchitis acute (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 0 | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Creatinine urine decreased (Investigations) | 0 | 1 | 1
Protein total decreased (Investigations) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 3 | 3
Partial seizures (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Angiokeratoma (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Diastolic hypertension (Vascular disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.